CLINICAL TRIAL: NCT06290271
Title: Correlation Between Changes in Arterial Wall Shear Stress and Prognosis Following Acute Major Intracranial Artery Occlusion and Recanalization
Brief Title: Arterial Wall Shear Stress After Intracranial Artery Recanalization
Status: Recruiting | Type: Observational
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Seoul National University Hospital (Other); Chungnam National University Hospital (Other); Asan Medical Center (Other); Chonnam National University Hospital (Other); Korea University Ansan Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Chan-Hyuk Lee, Prof., Ulsan University Hospital
Other Study IDs: CISTAR
Record Dates: First submitted 2023-11-02; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Intracranial Artery Occlusion
Keywords: Wall Shear Stress; Intracranial Artery Occlusion; Signal Intensity Gradient

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Passive Group: The cerebral blood flow pattern normalizes after the recanalization of the occluded artery
  Interventions: Other: Intracranial artery flow pattern
- Active Group: The overall major cerebral blood flow increases after the recanalization of the occluded artery
  Interventions: Other: Intracranial artery flow pattern

INTERVENTIONS:
Other: Intracranial artery flow pattern — the cerebral blood flow patterns observed after the occluded artery has been recanalized.

SUMMARY:
There has been consistent research on the cerebral blood flow features in ischemic stroke patients with acute occlusion of major intracranial arteries. However, studies analyzing the overall features of the major intracranial artery blood flow in the periods of pre and post-recanalization are still lacking. Time-of-flight magnetic resonance angiography (TOF-MRA) is extensively utilized to evaluate the intracranial arteries. The arterial signal intensity from MRA-TOF varies across subjects and arterial subtypes, leading to the development of the Signal Intensity Gradient (SIG) concept. SIG has demonstrated a strong correlation with Computational Fluid Dynamics (CFD), a known method for reflecting wall shear stress. SIG could be associated with the pathophysiology of wall shear stress. We aim to investigate the blood flow patterns and characteristics in the periods of pre and post-recanalization using SIG.

DETAILED DESCRIPTION:
1. Background The prognosis for ischemic stroke patients experiencing acute major intracranial artery occlusion is determined by a variety of factors. The status of arterial recanalization and the time taken to achieve recanalization play pivotal roles in determining patient outcomes. Even under similar conditions, short or long-term outcomes significantly differ among patients, making it challenging to solely explain with traditional risk factors. An acute occlusion in a major intracranial artery results in significant alterations in cerebral blood flow, enhancing flow through the Circle of Willis and collateral circulation to make up for the reduced blood supply to the affected area. After thrombectomy, the patterns of intracranial blood flow. changes again.

   Wall Shear Stress (WSS) is the frictional resistance force exerted by blood flow as it directly interacts with the vascular walls, and it serves as a critical indicator of vascular health. WSS is well-known for its correlation with atherosclerotic changes. Studies have shown that WSS in the internal carotid artery of ischemic stroke patients is lower compared to healthy individuals. Additionally, WSS was found to be reduced in the carotid artery of patients with lacunar infarctions. WSS in large artery strokes was lower than in the cardioembolic group. There have also been reports linking WSS to the progression of Moyamoya disease, suggesting that WSS may be associated with various vascular pathophysiologies, not just atherosclerotic changes.

   Time-of-Flight Magnetic Resonance Angiography (TOF-MRA) is a commonly used brain MRI technique, often utilized in conjunction with CT angiography to assess the course and condition of intracranial arteries. The signal intensity from MRA-TOF presents diverse distributions across different subjects and arteries. Based on this, the concept of Signal Intensity Gradient (SIG) has been derived. SIG has shown a strong correlation (correlation coefficient >0.8) with Computational Fluid Dynamics (CFD), a well-known method for assessing blood shear stress. In patients with the large artery atherosclerosis subtype of stroke, the SIG in the ipsilateral internal carotid artery was significantly lower than that on the contralateral side. These findings suggest a potential association between SIG, vascular shear stress, and the related pathophysiology.

   There is no need for additional imaging beyond TOF, and it is possible to measure even arteries of relatively small diameter. Therefore, SIG enables the analysis of shear stress pattern in major cerebral arteries before and after recanalization.
2. Aims We aim to investigate the blood flow patterns and characteristics in the periods of pre and post-recanalization using SIG.
3. Target number of participants A total of 160 participants (20 individuals from each center, total 8 centers)
4. Sample size assessment Although there haven't been many similar studies in the past, a study (PLoS One. 2020 Sep 21;15(9):e0238620) conducted a hemodynamic evaluation before and after major vessel recanalization, analyzing 11 patients. Sample size estimation using G*Power indicated that registration of approximately 144 patients would be necessary. Taking into account factors such as image quality, we anticipate an additional recruitment of about 10%, resulting in a final target of 160 cases.
5. Data Acquisition This study is a retrospective cohort study that involves the collection of electronic medical records and imaging data.

   Imaging Data to be Collected: (All images will be collected as DICOM files)
   * Brain MRI (Specific imaging conditions: Fluid Attenuated Inversion Recovery, Susceptibility Weighted Imaging, T1-Weighted Imaging, T2-Weighted Imaging, Diffusion Weighted Imaging, Apparent Diffusion Coefficient)
   * Brain MRA (Specific imaging conditions: source images from both extra and intracranial TOF-MRA, and 3D TOF-MRA)
6. Derivation of Intravascular Shear Stress (SIG) Through Image Analysis The transferred DICOM files are reconstructed into 3D vasculature using a separate software (VINT).

   SIG values for the major arterial segments within the cranial cavity are extracted.

   The major arterial segments are as follows, and the points where laminar flow of blood is formed were selected, considering the characteristics of the SIG technique:
   * Internal Carotid Artery: C1 distal segment prior to the horizontal intrapetrous segment
   * Vertebral Artery: V4 distal segment just before the formation of the basilar artery
   * Basilar Artery: mid to distal segment
   * Middle and Anterior Cerebral Arteries: proximal 1/2 or 1/3 segment
   * Posterior Cerebral Artery: P2 segment distal to the posterior communicating artery The measurements can be calculated into various SIG values (average, maximum, minimum, deviation).
7. Statistical Analysis Each patient will be classified into two groups based on their blood flow characteristics before and after recanalization. In a preliminary study, two types of blood flow (shear stress) changes were observed. Firstly, there was a pattern in which, following cerebral vascular occlusion, blood flow to the ischemic area was provided, and upon recanalization, it returned to the typical blood flow pattern. Secondly, there was a case where the overall blood flow in the major cerebral vessels increased after recanalization. To analyze these patterns, Paired t-test and Wilcoxon Signed-Rank Test will be used. (While this study is expected to proceed in the same manner as the group classification in the preliminary study, the classification method may be revised as the research progresses.)

For comparing mean values between groups, Independent Samples t-Test and Mann-Whitney U Test will be utilized. Categorical variables will be analyzed using the Chi-square Test or Fisher's Exact Test. Variables such as mRS (modified Rankin Scale), which are ordinal, will be assessed using the Mann-Whitney U Test or Wilcoxon Rank-Sum Test to utilize the median values.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and above
* Presenting with acute neurological impairments and demonstrating occlusion of major cerebral arteries (inclusive of one or more of the internal carotid artery, anterior cerebral artery, middle cerebral artery, posterior cerebral artery, vertebral artery, or basilar artery) as evidenced by brain MRA examinations
* Arterial recanalization subsequent to interventions such as intravenous thrombolysis and/or endovascular thrombectomy.
* Verification of the recanalized arteries on subsequent brain MRA imging
* Availability of source images from intracranial TOF-MRA (stored in DICOM format) both before and after arterial recanalization

Exclusion Criteria:

* Absence of TOF-MRA imaging either before or after arterial recanalization
* Brain MRI was performed, but TOF-MRA (DICOM source images) are missing
* Image analysis is deemed challenging due to the quality of the Brain MR images
* Intervention for vascular recanalization was unsuccessful, or re-occlusion was observed in the follow-up brain MRA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented to a medical center with acute neurological deficits and were confirmed to have acute occlusion in a major cerebral artery.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Neurological Severity at discharge | The Modified Rankin Scale (mRS) was assessed on the 7th day after admission.
  Modified Rankin Scale (mRS, 0-5, higher scores mean a worse outcome) measured at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Hwa Jung, Prof., Principal Investigator — Seoul National University Hospital; Hee Jung Song, Prof., Principal Investigator — Chungnam National University Hospital
Locations (8):
- South Korea (8):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ulsan University Hospital, Ulsan